CLINICAL TRIAL: NCT06950411
Title: Functionality Assessment of RadiSpine, an Artificial Intelligence Software as Medical Device for Lumbar Spine Quantification System
Brief Title: Validation of AI Lumbar Spine Anatomy Measureing Function
Acronym: Spinal cord
Status: Completed | Type: Observational
Sponsor: RadiRad Co., Ltd. (Industry)
Collaborators: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Sponsor
Other Study IDs: Validation of Spinal Anatomy
Record Dates: First submitted 2025-04-10; First posted 2025-04-30 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Spinal Cord Compression
Keywords: Artificial Intelligence(AI) Algorithm Spinal anatomy
MeSH Terms: conditions — Spinal Cord Compression

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Spinal degeneration and its associated clinical diseases are common ailments in aging societies. With the advent of a super-aging society, the importance of assistive technologies for spinal image interpretation is increasingly significant to enhance care efficiency and reduce medical personnel expenditure. Recently, due to the rapid development of artificial intelligence (AI) algorithm, AI-based computer-assisted detection (CADe) devices gradiually become a convenient method for spinal anatomy measurement. However, the accuracy of these devices has not been fully established. This study aims to validate the performance of RadiSpine (an application program) in spinal anatomy segmentation and measurement.

ELIGIBILITY:
Inclusion Criteria:

The subjects should be aged 20 or older and younger than 75, with an equal gender distribution of 50% male and 50% female. From this group, 150 subjects with reasonable datavalues will be selected, with a requirement that at least 30% of them are male and at least 30% are female.

Exclusion Criteria:

1. With history of spinal surgery
2. Spinal trauma
3. Spinal osteoporosis
4. Spinal metastasis or infection

Ages: 22 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The subjects should be aged 20 or older and younger than 75, with an equal gender distribution of 50% male and 50% female. From this group, 150 subjects with reasonable datavalues will be selected, with a requirement that at least 30% of them are male and at least 30% are female.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2024-09-12 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2025-03-31 (Actual)

PRIMARY OUTCOMES:
Segmentation accuracy (Mean) | 30 mins per individual
  The minimum Mean Dice Coefficient (MDC), defined as the lower limit of the 95% confidence interval (CI) for MDC, is above a predetermined allowable limit equal to 0.8

SECONDARY OUTCOMES:
Measurement accuracy | 30 mins per individual
  The maximum Mean Absolute Error (MAE), defined as the upper limit of the 95% CI for MAE, is below a predetermined allowable error limit equal to 2 mm

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei Veterans General Hospital, Taipei, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No